CLINICAL TRIAL: NCT01962337
Title: A Phase 1, Randomized, Double Blind, Placebo Controlled, Single and Multiple Ascending Dose Study of FPA008 in Healthy Volunteers and Subjects With Rheumatoid Arthritis
Brief Title: Phase 1 Single and Multiple Dose Study of FPA008 in Healthy Volunteers and Rheumatoid Arthritis Subjects
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: We have discontinued development of FPA008 in RA
Sponsor: Five Prime Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FPA008-001; 2013-003337-15 (EudraCT Number)
Record Dates: First submitted 2013-10-10; First posted 2013-10-14 (Estimated); Last update posted 2021-12-13 (Actual); Status verified 2021-12

CONDITIONS: Healthy; Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1-FPA008/Placebo Randomize DoseLevels1-4 (Experimental): Single infusion at 4 different dose levels
  Interventions: Drug: FPA008; Drug: Placebo
- 2-FPA008/Placebo Randomize DoseLevels1-2 (Experimental): Dual Infusions at 2 different dose levels
  Interventions: Drug: FPA008; Drug: Placebo
- 3-FPA008 Open-Label DoseLevels 1-3 (Experimental): Dual infusions at 1 dose level AND Dual/Triple infusions at 2 different dose levels
  Interventions: Drug: FPA008

INTERVENTIONS:
Drug: FPA008 — Infusion
Drug: Placebo — Infusion
  Arms: 1-FPA008/Placebo Randomize DoseLevels1-4; 2-FPA008/Placebo Randomize DoseLevels1-2

SUMMARY:
This is a Phase 1, randomized, double-blind, placebo-controlled study designed in 3 parts to assess the safety, tolerability, and PK of single and multiple ascending doses of FPA008 in adult healthy volunteers (Parts 1 and 2) and adult subjects with active RA (Part 3).

DETAILED DESCRIPTION:
Approximately 56 healthy volunteers will be enrolled at 1 study center in the Netherlands for Parts 1 and 2, and approximately 39 subjects will be enrolled at up to 6 sites in Central and Eastern Europe for Part 3. Dose escalations in Parts 1 and 2 will be driven by an assessment of the safety profile. Review of safety and PK parameters may inform decisions to add cohorts with intermediate dose levels in order to reach an optimal target exposure.

ELIGIBILITY:
Inclusion Criteria:

Part 1 and 2:

* Healthy adult male and female subjects between the ages of 21-55 years inclusive.
* Subject must be willing to remain in the Clinical Research Unit (CRU) for a minimum of 72 hours after each dose.

Part 3:

* RA male and female subjects between the ages of 21-70 years inclusive
* Evidence of active RA disease
* Inadequate response to biologic or non-biologic DMARDs
* Subjects will be required to be on background therapy with methotrexate.

Exclusion Criteria:

Parts 1, 2 and 3:

* BMI <18 or >32 kg/m2
* Clinically significant findings in physical exams and laboratory tests at screening and/or baseline
* Unwilling to abstain from alcohol for 48 hours prior to study start, during CRU confinement, as applicable, and for 48 hours prior to study visits.
* Unwilling to abstain from exercise more strenuous than walking during CRU confinement, as applicable, and for 48 hours prior to study visits.

Parts 1 and 2:

* Use of any prescription, non-prescription, or herbal medications as well as supplements or vitamins within 4 weeks prior to dosing, unless approved by the Investigator.
* Smoking more than 10 cigarettes, or the equivalent, per day.

Part 3:

* Current or previous history of inflammatory joint disease other than RA
* Evidence of extra-articular RA disease or systemic involvement
* Currently taking any medications other than those allowed per protocol guidelines
* Any surgical procedure including bone or joint surgery within 12 weeks prior to dosing
* Use of intra-articular (IA), intramuscular (IM), or IV corticosteroids for RA
* Neuropathies and neurovasculopathies
* Concomitant use of statins while on study.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2013-10; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events and dose-limiting toxicities of FPA008 administered in healthy volunteers and RA subjects | within 4-12 weeks
  Incidence of all-grade adverse events and dose limiting toxicities (DLT) during the DLT observation period and/or study treatment periods

CONTACTS AND LOCATIONS:
Overall Officials: Medical Lead, Study Director — Five Prime Therapeutics
Locations (6):
- Hungary (3):
  - BIK-Betegápoló Irgalmas rend-Budai Irgalmasrendi Kórház/Polyclinic of the Hospitaller Brothers of St. John of God in Budapest, Budapest
  - PRA Clinical Unit, Budapest
  - Drug Research Center, Kaposvár
- PRA Early Development Services, Groningen, Netherlands
- Poland (2):
  - Oddział Kliniczny Kliniki Chorób Wewnętrznych Szpitala Uniwersyteckiego w Krakowie, Krakow
  - MedPolina, Poznan